CLINICAL TRIAL: NCT00891306
Title: An Open-label Study to Assess the Efficacy and Safety of Alipogene Tiparvovec (AMT-011), Human LPL [S447X], Expressed by an Adeno-Associated Viral Vector After Intramuscular Administration in LPL-deficient Adult Subjects
Brief Title: Efficacy and Safety of Human Lipoprotein Lipase (LPL)[S447X] Expressed by an Adeno-Associated Viral Vector in LPL-deficient Subjects
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amsterdam Molecular Therapeutics (Industry)
Collaborators: The Clinical Trial Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-AMT-011-02
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Familial Lipoprotein Lipase Deficiency
Keywords: LPLD, Lipoprotein Lipase Deficiency; Chylomicronemia; Gene therapy; AAV; Lipoprotein Lipase; Alipogene tiparvovec; AMT-011
MeSH Terms: conditions — Hyperlipoproteinemia Type I | interventions — Alipogene tiparvovec; Mycophenolic Acid; Cyclosporine; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Gene Therapy
  Interventions: Genetic: Alipogene Tiparvovec (AMT-011), Human LPL [S447X]; Drug: mycophenolate mofetil; Drug: cyclosporine; Drug: methylprednisolone

INTERVENTIONS:
Genetic: Alipogene Tiparvovec (AMT-011), Human LPL [S447X] — intra muscular, 1 x E12 gc per kg body weight, injected in a single series of intramuscular injections
  Other Names: Glybera; AMT-011
Drug: mycophenolate mofetil — oral, 2 g/day, day -3 till week 12
  Other Names: CellCept
Drug: cyclosporine — oral, 3 mg/kg/day, day -3 till week 12
  Other Names: Neoral
Drug: methylprednisolone — single intravenous bolus of methylprednisolone (1 mg/kg bodyweight)
  Other Names: Solumedrol®

SUMMARY:
This trial is designed to expand the currently available data on the safety and efficacy of alipogene tiparvovec treatment in lipoprotein lipase deficiency (LPLD) and to further the understanding of possible mechanisms of action of the therapy.

DETAILED DESCRIPTION:
LPLD is a rare autosomal recessive disorder, characterized by the presence of marked chylomicronemia and hence hypertriglyceridemia. Clinically the most severe manifestation of chylomicronemia, is acute pancreatitis, which can be lethal. There is no effective therapy available to modulate the course of the illness and prevent complications for these patients. The current clinical management consists of severe reduction of dietary fat that is hard if not almost impossible to comply with. LPLD subjects continue to experience pancreatitis attacks, and are admitted to intensive care units on several occasions.

Alipogene tiparvovec corrects or restores lipoprotein lipase (LPL) function long term, and hence reverses some symptoms, halts the disease progression and prevents further complications. Alipogene tiparvovec gene therapy ensures that a catabolically beneficial variant of the human LPL gene, LPL[S447X] is expressed and active in the relevant tissues in humans. Delivery of the gene is realized via intramuscular injection of an adeno-associated viral vector, pseudotyped with AAV1 capsids.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with LPLD defined as:

  * Confirmed homozygosity or compound heterozygosity for the mutations in the LPL gene, resulting in LPL deficiency
  * Having a post heparin plasma LPL activity of ≤ 20% of normal or a well defined mutation for which it is documented that the LPL mass and activity are within the limits described above
  * Having a history of pancreatitis
  * Having fluctuating TG concentrations with median fasting plasma TG concentrations > 10.00 mmol/L
* Being in good general physical health with, in the opinion of the investigator:

  * No other clinically significant and relevant abnormalities in the medical history which could interfere with the participation to the study
  * No clinically significant abnormalities at the physical examination which could interfere with the participation to the study
  * No clinically significant abnormalities at the routine laboratory evaluation performed prior to the trial
* Women of non-child bearing potential or with a negative pregnancy test.
* Non breast feeding women
* Women using appropriate contraceptive (if relevant) and their partner using barrier contraception 2 weeks before starting immunosuppressive therapy
* Men practicing barrier birth control and their partner using appropriate contraception.
* Willing to fully comply with all study procedures and requirements of the trial such as restrictions to a low-fat diet.

Exclusion Criteria:

* Having a chronic inflammatory muscle disease.
* Any current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may make the subject unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures based on the investigator's opinion(eg. malignant neoplasia)
* Active infectious disease of any nature, including clinically active viral infections
* Having one of the following outcomes from the blood screening tests after appropriate correction due to the presence of chylomicronemia:

  * Platelet count < 100 x 109 /L
  * Hemoglobin < 6.2 mmol/L
  * Liver function disturbances (bilirubin ≥1.5 x normal, ALT > 2 x ULN (upper limit of normal)
  * CPK > 2 x ULN
  * Cockcroft-Gault estimated creatinine clearance < 50cc/min
  * PT and PTT outside normal range or not determinable unless judged as acceptable for the subjects by the investigator
  * Having a positive test for HIV, Hepatitis B, Hepatitis C or being positive for tuberculosis
* Obesity defined as body mass index (BMI) > 30 kg/m2
* Having a recent history of alcohol or drug abuse e.g. barbiturates, cannabinoids and amphetamines, and the subject is positive in a urine screen for drugs of abuse
* Using anti-coagulants
* Participation in another clinical trial or receipt of any other investigational drug within 30 days of screening or planning to participate in another clinical trial during the course of the study, except observational studies
* Subjects which cannot be treated with immunosuppressive medication or steroids
* Known to be allergic to any constituent of the therapy (including the immune suppressors) or a having a condition that prohibits the use of therapy
* Received previous treatment with AMT-010, Alipogene tiparvovec or other gene therapy investigational product
* Requiring a post heparin plasma LPL activity test for diagnostic confirmation and having a history of heparin induced thrombocytopenia or other heparin related complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Reduction of triglyceride (TG) concentrations | 12 weeks

SECONDARY OUTCOMES:
Reduction of chylomicrons and/or chylomicron-TG ratio | 12 weeks
To determine the biological activity and expression of the lipoprotein lipase [LPLS447X] transgene product | 14 weeks
To assess the safety profile | 14 weeks
To assess shedding of viral vector | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gaudet, MD, Ph.D., Principal Investigator — ECOGENE-21 Clinical Trial Center / Centre de santé et de services sociaux de Chicoutimi, Chicoutimi Hospital, Quebec, Canada
Locations (2):
- Canada (2):
  - ECOGENE-21 Clinical Trial Center / Centre de santé et de services sociaux de Chicoutimi, Chicoutimi, Quebec
  - Centre des Maladies Lipidiques de Québec, Québec, Quebec

REFERENCES:
- [Background] Rip J, Nierman MC, Sierts JA, Petersen W, Van den Oever K, Van Raalte D, Ross CJ, Hayden MR, Bakker AC, Dijkhuizen P, Hermens WT, Twisk J, Stroes E, Kastelein JJ, Kuivenhoven JA, Meulenberg JM. Gene therapy for lipoprotein lipase deficiency: working toward clinical application. Hum Gene Ther. 2005 Nov;16(11):1276-86. doi: 10.1089/hum.2005.16.1276. PMID 16259561
- [Background] Ross CJ, Twisk J, Meulenberg JM, Liu G, van den Oever K, Moraal E, Hermens WT, Rip J, Kastelein JJ, Kuivenhoven JA, Hayden MR. Long-term correction of murine lipoprotein lipase deficiency with AAV1-mediated gene transfer of the naturally occurring LPL(S447X) beneficial mutation. Hum Gene Ther. 2004 Sep;15(9):906-19. doi: 10.1089/hum.2004.15.906. PMID 15353045
- [Background] Ross CJ, Liu G, Kuivenhoven JA, Twisk J, Rip J, van Dop W, Excoffon KJ, Lewis SM, Kastelein JJ, Hayden MR. Complete rescue of lipoprotein lipase-deficient mice by somatic gene transfer of the naturally occurring LPLS447X beneficial mutation. Arterioscler Thromb Vasc Biol. 2005 Oct;25(10):2143-50. doi: 10.1161/01.ATV.0000176971.27302.b0. Epub 2005 Jul 7. PMID 16002740
- [Background] Ross CJ, Twisk J, Bakker AC, Miao F, Verbart D, Rip J, Godbey T, Dijkhuizen P, Hermens WT, Kastelein JJ, Kuivenhoven JA, Meulenberg JM, Hayden MR. Correction of feline lipoprotein lipase deficiency with adeno-associated virus serotype 1-mediated gene transfer of the lipoprotein lipase S447X beneficial mutation. Hum Gene Ther. 2006 May;17(5):487-99. doi: 10.1089/hum.2006.17.487. PMID 16716106
- [Background] Stroes ES, Nierman MC, Meulenberg JJ, Franssen R, Twisk J, Henny CP, Maas MM, Zwinderman AH, Ross C, Aronica E, High KA, Levi MM, Hayden MR, Kastelein JJ, Kuivenhoven JA. Intramuscular administration of AAV1-lipoprotein lipase S447X lowers triglycerides in lipoprotein lipase-deficient patients. Arterioscler Thromb Vasc Biol. 2008 Dec;28(12):2303-4. doi: 10.1161/ATVBAHA.108.175620. Epub 2008 Sep 18. No abstract available. PMID 18802015
- [Derived] Carpentier AC, Frisch F, Labbe SM, Gagnon R, de Wal J, Greentree S, Petry H, Twisk J, Brisson D, Gaudet D. Effect of alipogene tiparvovec (AAV1-LPL(S447X)) on postprandial chylomicron metabolism in lipoprotein lipase-deficient patients. J Clin Endocrinol Metab. 2012 May;97(5):1635-44. doi: 10.1210/jc.2011-3002. Epub 2012 Mar 21. PMID 22438229
- See also: Related Info — http://www.amtbiopharma.com/